CLINICAL TRIAL: NCT02437370
Title: Feasibility Trial of MK3475 + Docetaxel or Gemcitabine in Platinum Pre-treated Urothelial Cancer
Brief Title: Pembrolizumab and Docetaxel or Gemcitabine Hydrochloride in Treating Patients Urothelial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 723260; UCDCC#252 (Other: UC Davis); UCDCC#252 (Other: University of California Davis Comprehensive Cancer Center); 51521 (Other Grant/Funding Number: Merck); NCI-2015-00426 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Urothelial Carcinoma of the Renal Pelvis and Ureter; Recurrent Bladder Carcinoma; Recurrent Urothelial Carcinoma of the Renal Pelvis and Ureter; Regional Urothelial Carcinoma of the Renal Pelvis and Ureter; Stage III Bladder Urothelial Carcinoma; Stage III Urethral Cancer; Stage IV Bladder Urothelial Carcinoma; Stage IV Urethral Cancer; Urethral Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — pembrolizumab; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (pembrolizumab, docetaxel) (Experimental): pembrolizumab IV over 30 minutes on day 1 and docetaxel IV over 60 minutes on day 1.
  Interventions: Drug: Pembrolizumab; Drug: Docetaxel
- Arm B (pembrolizumab, gemcitabine hydrochloride) (Experimental): pembrolizumab IV as in Arm A and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8.
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Pembrolizumab — Given IV
  Other Names: Keytruda; MK-3475
Drug: Docetaxel — Given IV
  Arms: Arm A (pembrolizumab, docetaxel)
Drug: Gemcitabine Hydrochloride — Given IV
  Arms: Arm B (pembrolizumab, gemcitabine hydrochloride)

SUMMARY:
This phase I trial studies the side effects and best dose of pembrolizumab when given together with docetaxel or gemcitabine hydrochloride in treating patients with previously treated urothelial cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) or that has spread from the primary site (place where it started) to other places in the body (metastatic). Monoclonal antibodies, such as pembrolizumab, may block tumor growth in different ways by targeting certain cells. Drugs used in chemotherapy, such as docetaxel and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab together with docetaxel or gemcitabine hydrochloride may be a better treatment for urothelial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of MK-3475 (pembrolizumab) when given in combination with docetaxel or gemcitabine (gemcitabine hydrochloride) in patients with advanced or metastatic platinum-treated urothelial cancer.

SECONDARY OBJECTIVES:

I. To assess in a preliminary manner the efficacy of this combination (overall response rate and progression free survival).

II. To determine in an exploratory manner programmed death (PD)-ligand (L)1 expression in archival tumor specimens and to correlate this with patient outcomes.

OUTLINE: This is a dose-escalation study of pembrolizumab. Patients are assigned to 1 of 2 treatment arms. (Patients who had received prior gemcitabine hydrochloride/cisplatin or gemcitabine hydrochloride/carboplatin [GC] or methotrexate, vinblastine sulfate, adriamycin, and cisplatin [MVAC] therapy are assigned to Arm A).

ARM A: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and docetaxel IV over 60 minutes on day 1.

ARM B: Patients receive pembrolizumab IV as in Arm A and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8.

In both arms, treatment repeats every 21 days for 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Have locally advanced or metastatic urothelial cancer that is not amenable to curative surgical treatment

  * Have histologically or cytologically confirmed urothelial tract carcinoma
* Be previously chemotherapy-treated; all patients may have received up to two prior lines of chemotherapy (excludes systemic therapy) for recurrent/advanced disease, as long as one of those regimens was platinum-based; (it is anticipated that patients would have been previously treated with MVAC or GC, or variations of these standard frontline regimens)
* Be willing and able to provide written informed consent for the trial
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion
* Life expectancy of greater than 6 months
* Have a performance status of 0 to 1 on the Zubrod performance scale
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated* creatinine clearance >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN; (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl])

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Alkaline phosphatase not applicable (N/A)
* International normalized ratio (INR) or prothrombin time (PT) =<1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has known hypersensitivity to MK-3475 (pembrolizumab) or any of its incipients
* Patients with a known hypersensitivity to gemcitabine (Arm B only)
* Patients with hypersensitivity to docetaxel or polysorbate 80 (Arm A only)
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy; free of disease for more than 5 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment; anti-coagulants are permitted
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active serious bacterial infection requiring systemic antimicrobial therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cluster of differentiation (CD)137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of pembrolizumab based on the incidence of dose limiting toxicity, defined as the Incidence of adverse events, using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 6 months post-treatment
  Will be summarized descriptively by tables of numbers and percent of patients experiencing adverse events, overall and by type, grade, seriousness, duration, action taken, and assessment of relation to pembrolizumab or docetaxel or gemcitabine hydrochloride.

SECONDARY OUTCOMES:
Overall response rate (ORR), assessed using the RECIST version 1.1 | Up to 6 months post-treatment
  The number and proportion experiencing complete response, partial response, stable disease, or progressive disease will be summarized separately for each study arm.
Progression free survival (PFS) | Time from enrollment to the first occurrence of disease progression, as determined by RECIST v1.1, or death from any cause, assessed up to 6 months post-treatment
  Will be summarized graphically by Kaplan-Meier curves and descriptively by a corresponding life-table approach to allow for possible censored data.
PD-L1 expression | Baseline
  The relation of PD-L1 expression at baseline to outcome (ORR and PFS) will be summarized descriptively in exploratory analyses, separately for each study arm. Descriptive associations with ORR will be summarized by the means and standard deviations for responders vs. non-responders, and graphically by dot plots of PD-L1 expression for responders and non-responders. Descriptive associations with PFS will be summarized by Kaplan-Meier plots comparing PFS for high and low PD-L1 expression.

CONTACTS AND LOCATIONS:
Overall Officials: Primo Lara, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States